CLINICAL TRIAL: NCT03547193
Title: Evaluation of Two Neck Ultrasound Measurements as Predictors of Difficult Laryngoscopy: a Prospective Trial
Brief Title: Two Neck Ultrasound Measurements as Predictors of Difficult Laryngoscopy
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Study Director, Università Politecnica delle Marche
Other Study IDs: 2016-0405
Record Dates: First submitted 2018-05-12; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Anesthesia; Airway Complication of Anesthesia; Difficult Intubation
Keywords: difficult laringoscopy; difficult airway; airway management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Unpredictable laryngoscopic difficulty remains a dramatic challenge for anaesthesiologists. Ultrasound (US) based airway assessment has been recently proposed as a useful tool in adjunct to clinical methods, but to date few studies are available about the potential role of ultrasound in difficult airway evaluation.

The aim of this study is to determine the correlation between the sonographic measurements of anterior cervical soft tissues's thickness and Cormack-Lehane grade view at direct laryngoscopy in patients with normal clinical screening tests.

Design: Prospective, single blinded, observational study. Number of patients: 300 adult patients Methods: All patients are assessed before surgery to evaluate clinical evidence of difficult airways. Simultaneous ultrasound measures of the anterior cervical soft tissues are performed.

At induction of anaesthesia the laryngoscopic view is graded by a different anaesthetist, blinded to the ultrasound assessments.

Statistical analysis:

Receiver operating characteristic curves (ROC) are used to determine the "difficulty prediction capability" of each sonographic measurement and to assess the optimal cut-off scores To allow for comparisons between "restricted-difficult" airway and "easy" airway groups, a two-sided Student's t-test and Fisher's exact test is employed as appropriate. The results will be averaged (mean ± standard deviation SD) for each parameter for continuous data. Values of p < 0.05 are considered as statistically significant.

DETAILED DESCRIPTION:
Unpredictable laryngoscopic difficulty, especially if difficult ventilation occurs, during standard laryngoscopy, remains a dramatic challenge for anaesthesiologists. Accurate airway assessment should always be performed, but the common clinical screening tests have shown low sensitivity and specificity with a limited predictive value. Ultrasound (US) based airway assessment has been recently proposed as a useful, simple, bedside and non-invasive tool in adjunct to clinical methods, but to date few studies are available about the potential role of ultrasound in difficult airway evaluation and these are mostly limited on specific groups of patients.

The aim of this prospective, single blinded, observational study is to determine the correlation between two neck ultrasound measures assessed at the pre-operative visit and Cormack-Lehane grade view at direct laryngoscopy, assessed at the induction of anaesthesia 24 hours later.

METHODS: During the pre-operative visit (24 hours before surgery), clinical screening tests to predict a difficult airway are performed and the anterior cervical soft tissue's thickness is assesses.

The thickness of the anterior cervical soft tissues is measured at two levels, thyro-hyoid membrane (pre-epiglottis space) and vocal cords (laryngeal inlet), using a US probe 10-13-MHz linear transducer placed in the transverse plane with the patient's head in neutral position.

On each level the distance from the skin in the median axis in cm (mDSE = median distance skin to epiglottis; mVC = median distance skin to vocal cords) and the surrounding Area in cm2 (PEA = pre-epiglottis area; AVC = Area pre vocal cords) are measured.

At the induction of anaesthesia the laryngoscopic view is graded by a different anaesthetist blinded to the ultrasound assessments and with more than 5 years of experience with OR activity. For each patient it's considered only the best attempt at direct laryngoscopy obtained after optimizing position, complete muscle relaxation (TOF=0), and, if necessary, external laryngeal manipulation. A decrease of SpO2 < 92% is a criterion for abandoning the procedure and a maximum of three attempts are admitted before declaring intubation failure with direct laryngoscopy. A Cormack-Lehane Grade 1 or 2a are classified as easy laryngoscopy and grade 2b - 3a - 3b or 4 as restricted or difficult laryngoscopy.

STATISTICAL ANALISYS: According to the literature, ultrasound measurements should predict as difficult at least 80% of the intubations that are really difficult (with a C-L ≥ 2b). Since the incidence of difficult intubation is about 5-10% of all intubations 1-3,6, it is necessary to study at least 244 patients in order to obtain statistically significant differences between the two groups accepting an alpha error of 0.05 and a beta error of 0.20.

Kolmogorov-Smirnov's test is used to test the normality of distribution. Receiver operating characteristic curves (ROC) is used to determine the "difficulty prediction capability" of each sonographic measurement and to assess the optimal cut-off scores To allow for comparisons between "restricted-difficult" airway and "easy" airway groups, a two-sided Student's t-test and Fisher's exact test are employed as appropriate. The results will be averaged (mean ± standard deviation SD) for each parameter for continuous data. Values of p < 0.05 were considered as statistically significant.

ETHICS: Ethical approval for this study was provided by Marche's Regional Ethics Committee (CERM), Ancona, ITA (Protocol No. 2016-0405); Chairperson: Prof Marcello D'Errico on 23 March 2017. Informed written consent was obtained. The study conformed to the Declaration of Helsinki and Good Clinical Practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing pre-operative evaluation for elective surgery

Exclusion Criteria:

* Predicted difficult intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the adult patients undergoing to pre-operative evaluation for elective surgery at AOU-University Hospital of Ancona
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
median Distance Skin to Epiglottis (mDSE) | 24 hours
  The median Distance Skin to Epiglottis, unit of measure cm, is detected using a US linear probe (10-13-MHz) with the transducer placed in the transverse plane and the patient's head in neutral position. It represents the distance from the skin in the median axis and the epiglottis

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, MD, PhD, Study Director — UNIVPM, University of Ancona
Locations (1):
- AOU Ospedali Riuniti Ancona - Università Politecnica delle Marche, Ancona, Italy

REFERENCES:
- [Derived] Falcetta S, Cavallo S, Gabbanelli V, Pelaia P, Sorbello M, Zdravkovic I, Donati A. Evaluation of two neck ultrasound measurements as predictors of difficult direct laryngoscopy: A prospective observational study. Eur J Anaesthesiol. 2018 Aug;35(8):605-612. doi: 10.1097/EJA.0000000000000832. PMID 29889671